CLINICAL TRIAL: NCT06924242
Title: Thyroid Cancer in Surgically Treated Multinodular Goiter: Incidence and Histopatological Outcomes
Brief Title: Thyroid Cancer in Surgical Treated Multinodular Goiter
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Giovanna Pavone, Medical Doctor, University of Foggia
Other Study IDs: 10
Record Dates: First submitted 2025-03-28; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Goiter, Nodular; Total Thyroidectomy; Thyroid Cancer
MeSH Terms: conditions — Goiter, Nodular; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with multinodular goiter who underwent total or partial thyroidectomy
  Interventions: Procedure: total or partial thyroidectomy

INTERVENTIONS:
Procedure: total or partial thyroidectomy — Total thyroidectomy is a surgical procedure that involves the complete removal of the thyroid gland. It is performed to treat conditions such as thyroid cancer, large goiters, or severe hyperthyroidism. The surgery is typically conducted under general anesthesia through an incision in the lower neck. Postoperative management may include hormone replacement therapy with levothyroxine to compensate for the loss of thyroid function. Potential complications include hypocalcemia due to parathyroid gland injury and vocal cord dysfunction from recurrent laryngeal nerve damage.

SUMMARY:
This study aims to investigate, based on existing knowledge, the incidence of occult thyroid carcinoma in a cohort of patients with MNG, providing new insights into the prevalence and characteristics of thyroid malignancies in MNG. It seeks to contribute to optimizing diagnostic evaluations for patients with multinodular goiter.

DETAILED DESCRIPTION:
This retrospective study included patients with a preoperative diagnosis of multinodular goiter who underwent total or partial thyroidectomy from January 2018 to May 2024 at the Department of Medical and Surgical Sciences at the University Hospital "Ospedali Riuniti" in Foggia. The study's objective was to investigate the incidence of thyroid carcinoma in patients undergoing thyroidectomy for MNG, also analyzing associated demographic and clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with multinodular goiter via thyroid ultrasound, with or without FNA cytology.
* patients who underwent surgery.
* availability of complete clinical data

Exclusion Criteria:

* history of thyroid carcinoma or other thyroid neoplasms.
* not completed postoperative follow up.
* patients with preoperative FNA results indicating malignancy (TIR 4-5), suspicion of malignancy (TIR 3), or indeterminate significance (TIR 1)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of both sex with cancer incidence in multinodular thyroid goiter who underwent surgery in the same center
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
incidence of occult thyroid carcinoma | 6 years
  Incidence of occult thyroid carcinoma in a cohort of patients with multinodular goiter, providing new insights into the prevalence and characteristics of thyroid malignancies.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Foggia, Foggia, FG, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT06924242/Prot_000.pdf